CLINICAL TRIAL: NCT02827188
Title: Cognitive Restructuring in ADHD: Functional Training
Acronym: CRAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Ehave (Other); Ontario Brain Institute (Other)
Responsible Party: Principal Investigator, Jennifer Crosbie, Psychologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB1000045526
Record Dates: First submitted 2016-05-09; First posted 2016-07-11 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Attention-deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Subjects randomly assigned to this arm will train on the Mega Team video game.
  Interventions: Other: Mega Team-videogame
- Control-waitlist group (No Intervention): Subjects randomly assigned to this arm will be the wait-list group. They are allowed to play the video games that they usually play.

INTERVENTIONS:
Other: Mega Team-videogame — Subjects randomly assigned to the treatment group will be instructed to practice Mega Team for 30-35 minutes a day, approximately 5 days a week for a minimum of 21 days and a maximum of 25 days.
  Other Names: Mega Team
  Arms: Treatment group

SUMMARY:
The objective of the Cognitive Restructuring in ADHD: Functional Training (CRAFT) study is to develop a non-pharmacological intervention program for children with Attention Deficit Hyperactivity Disorder (ADHD). ADHD is a childhood onset clinical disorder of inattention, hyperactivity, and impulsivity. The present study will investigate the validity, feasibility and efficacy of this novel intervention.

DETAILED DESCRIPTION:
This study will consist of a pre-post design and will include three phases. Participants will be tested individually at SickKids at baseline and post-training, the training phase will take place at the participants' respective homes. Each participant's parent will complete a demographic/medical questionnaire. The cognitive and behavioural outcome measures of interest in this study will be the following:

Planning and Organization: Tower Test from the Delis-Kaplan Executive Function System (D-KEFS; Delis et al, 2001) is a test of planning and problem solving abilities. Participants are asked to construct towers of discs on a set of pegs corresponding to a model. Raw scores reflect the participant's ability to use the fewest possible moves to achieve the tower depicted in the model.

Response Inhibition: Inhibitory control will be measured using the Stop Signal Task (SST). The SST measures the ability to cancel an already initiated motor response. The primary outcome measure will be the participants' mean stop signal reaction time (SSRT).

Inattentive and Hyperactivity Behaviour: Items associated with inattentiveness and hyperactivity from the Swanson, Nolan and Pelham Teacher and Parent Rating Scale version 4 (SNAP IV) will be used to estimate behavioural symptoms associated with ADHD.

Academic Performance: Academic efficiency and accuracy will be assessed using the fluency measures from the Woodcock Johnson III (WJ III) test of achievement.

Spatial Span: The spatial span item from the Wechsler Intelligence Scale for Children (WISC) will be used to estimate the child's visuo-spatial span. The primary outcome measure will be the number of correctly recalled spatial locations.

Working Memory: Working Memory will be tested using Spatial N-back 0,1,2.

Phase 1: Baseline Session

Children and their parents will participate in a 2 hour clinic session at SickKids. During this appointment, investigator/research staff will assess children's cognitive performances. The cognitive measures have been selected based on the range of processes commonly impaired in children with ADHD which will also be targeted by Mega Team. Both the training group and the control group will complete the same assessment battery. Tasks and questionnaires that will be included in this battery are;

* Spatial Span (working memory)
* WJ III
* Tower Test (D-KEFS)
* SST
* SNAP
* Demographic/Medical questionnaire
* Spatial N-back 0,1,2

Spatial Working Memory has been shown to be impaired in ADHD. In this task, the experimenter will point to a sequence of spatial locations on a grid and children will be required to reproduce this sequence in a forward or backward order. The length of sequences will vary between sets of 2-7. The spatial span tasks will be scored based on the Spatial Span scoring rules and norms (WISC-IV Integrated).

Academic efficiency and accuracy will be assessed using the fluency measures from the Woodcock Johnson III (WJ III) test of achievement. Participants will complete the reading fluency, math fluency and writing fluency subtests using alternate forms A and B in each assessment period to prevent retesting bias. This battery has been selected to be included in this study to provide objective measures of academic performance in areas where children with ADHD often show weakness (Czamara et al., 2013, Greven et al.,2013, Schmiedeler and Schneider, 2013).

Tower Test (DKEFS subtest (Delis et al., 2001) is a test of planning and problem solving abilities. Planning and organizational deficits have been reported in children with ADHD (Grodzinsky and Diamond, 1992, Mataro et al., 1997, Wilcutt et al., 2005) and will be targeted by Mega Team. Participants will be asked to construct towers of discs on a set of pegs corresponding to a model. Raw scores reflecting the participant's ability to use the fewest possible moves to achieve the tower depicted in the model.

The Stop Signal Test (SST) is a measure of response inhibition. Difficulties of response inhibition in ADHD have been reported by 82% of studies that have examined it. Response inhibition has been posited as an endophenotype for ADHD and shown to distinguish a group of children with ADHD from one with ADHD symptoms and one with conduct disorder. In the SST, participants will perform a choice reaction time task and will be instructed to respond as quickly and accurately as possible. On a portion of trials (e.g. 25%) a stop signal (a tone) will be presented and participants will be required to restrain their motor response. The delay between the go stimulus (the primary task) and the onset of the stop signal varies to determine the participant's ability to stop an already initiated motor response. This individualized stopping latency varies as a function of impulsivity. The stop-signal reaction time (SSRT) provides a measure of the ability to inhibit an already initiated response.

The SNAP-IV parent 18-item Rating Scale is a standardized scale that measures symptoms associated with ADHD. This provides the opportunity to identify the child's behavioural issues relative to standardized norms. This measure includes the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criteria for ADHD with items 1-9 representing the inattentive subset of symptoms and items 10-18 representing the Hyperactivity/Impulsivity subset. Parents will be requested to fill out this scale at baseline, during training and post-training.

Spatial N-back 0,1,2 - The N-Back task requires on-line monitoring, updating, and manipulation of remembered information and measures key processes within working memory. In the N-Back task, the participant is required to monitor a series of stimuli and to respond whenever a stimulus is presented that is the same as the one presented n trials previously, where n is a pre-specified integer, usually 0, 1, or 2. The current study will use spatial location (spatial) paradigms.

Phase 2: the Training Sessions

In this phase, children in the treatment group will train at home on a computer with internet connection. They will be instructed to practice Mega Team for 30-35 minutes a day, approximately 5 days a week for a minimum of 21 sessions and a maximum of 25 sessions. The minimum value of 21 sessions has been selected based on findings of prior research. Majority of studies have been able to capture significant training-induced improvements after 21 sessions. The maximum training session of 25 days has been set to control for variability within and between our groups.

Performance on Mega Team will automatically upload to a secure website which will be monitored by the experimenters for both compliance and data analyses purposes. For example, research staff will know how often and how long the participants trained on Mega Team. One of the major objective of this study is to design a training program that is inherently engaging to children so that it will be easier to comply with the training schedule. It is possible that the presence of certain comorbid conditions such as ODD will affect adherence. However, the goal is to avoid compliance issues by ensuring that Mega Team is game-like and interesting to all children.

Children in the control group will play video-games as usual. Participants' parent/guardian in both groups (Treatment, Control) will be asked to complete a video game usage log weekly to record the type and duration of video game playing. Parents of both groups will also be required to fill out the SNAP-IV parent 18-item questionnaire once a week during the training phase. This questionnaire will provide a measure of change in behaviour.

Phase 3: the Post-Training Session

Following the completion of the training, families from both the treatment and the control groups will be scheduled for another 2 hour clinic session. The time between the completion of training and post-training appointment will range between 2-7 days. At this appointment, families will be asked to complete the same tasks and questionnaires that were administered to them during the baseline session. In this session, children will also be asked to fill out the Video-game Questionnaire. At the end of the post-training visit participants in the control group will be sent home with access to the Mega Team game for the same duration as the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 6-12 years old
* Subject has a diagnosis of Attention Deficit Hyperactive Disorder
* Subject is a previous POND baseline study (Attention Deficit Hyperactive Disorder Cognitive deficit and syndrome definition) participant.
* Parent/legal guardian and subject are willing to consent/assent to participate in this study

Exclusion Criteria:

* IQ below 80 on both verbal and performance scales of the Wechsler Intelligence Scale for children (WISC)-IV/V or Wechsler Abbreviated scale of intelligence (WASI II)
* History of psychosis, schizophrenia or other major mental health diagnosis that will prevent participation/completion of the protocol
* Subject's current medical problems that would preclude his/her participation in the study
* Child younger than 6 years old or older than 12
* Parent/legal guardian and/or subject not willing to consent/assent to participate in this study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

PRIMARY OUTCOMES:
Change in Response inhibition | Baseline and post-training study visits (4-5 weeks apart)
  Inhibitory control will be measured using the Stop Signal Task.
Change in Working memory | Baseline and post-training study visits (4-5 weeks apart)
  Target accuracy as measured by the N-Back Tasks

SECONDARY OUTCOMES:
Change in Inattentive and Hyperactivity Behaviour | Baseline, week1, week 2, week 3, week 4, and at post-training study visit (week 4-5)
  Measured by SNAP IV
Change in Planning and Organization | Baseline and post-training study visits (4-5 weeks apart)
  will be measured using the Tower Test from the Delis-Kaplan Executive Function System
Change in Academic performance | Baseline and post-training study visits (4-5 weeks apart)
  Academic efficiency and accuracy will be assessed using the fluency measures from the Woodcock Johnson III (WJ III) test of achievement
Change in Spatial Span | Baseline and post-training study visits (4-5 weeks apart)
  We will use the spatial span item from the WISC to estimate the child's visuo-spatial span

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Crosbie, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be shared with our sponsor/funders- Ontario Brain Institute and ehave.

REFERENCES:
- [Background] Chein JM, Morrison AB. Expanding the mind's workspace: training and transfer effects with a complex working memory span task. Psychon Bull Rev. 2010 Apr;17(2):193-9. doi: 10.3758/PBR.17.2.193. PMID 20382919
- [Background] Crosbie J, Perusse D, Barr CL, Schachar RJ. Validating psychiatric endophenotypes: inhibitory control and attention deficit hyperactivity disorder. Neurosci Biobehav Rev. 2008;32(1):40-55. doi: 10.1016/j.neubiorev.2007.05.002. Epub 2007 May 18. PMID 17976721
- [Background] Czamara D, Tiesler CM, Kohlbock G, Berdel D, Hoffmann B, Bauer CP, Koletzko S, Schaaf B, Lehmann I, Herbarth O, von Berg A, Muller-Myhsok B, Schulte-Korne G, Heinrich J. Children with ADHD symptoms have a higher risk for reading, spelling and math difficulties in the GINIplus and LISAplus cohort studies. PLoS One. 2013 May 27;8(5):e63859. doi: 10.1371/journal.pone.0063859. Print 2013. PMID 23724008
- [Background] Dahlin E, Nyberg L, Backman L, Neely AS. Plasticity of executive functioning in young and older adults: immediate training gains, transfer, and long-term maintenance. Psychol Aging. 2008 Dec;23(4):720-30. doi: 10.1037/a0014296. PMID 19140643
- [Background] Greven CU, Kovas Y, Willcutt EG, Petrill SA, Plomin R. Evidence for shared genetic risk between ADHD symptoms and reduced mathematics ability: a twin study. J Child Psychol Psychiatry. 2014 Jan;55(1):39-48. doi: 10.1111/jcpp.12090. Epub 2013 Jun 3. PMID 23731013
- [Background] Hazel-Fernandez LA, Klorman R, Wallace JM, Cook S. Methylphenidate improves aspects of executive function in African American children with ADHD. J Atten Disord. 2006 May;9(4):582-9. doi: 10.1177/1087054705284243. PMID 16648225
- [Background] Schmiedeler S, Schneider W. Attention-deficit hyperactivity disorder (ADHD) in the early years: diagnostic issues and educational relevance. Clin Child Psychol Psychiatry. 2014 Jul;19(3):460-75. doi: 10.1177/1359104513489979. Epub 2013 Jun 19. PMID 23785052
- [Background] Shue KL, Douglas VI. Attention deficit hyperactivity disorder and the frontal lobe syndrome. Brain Cogn. 1992 Sep;20(1):104-24. doi: 10.1016/0278-2626(92)90064-s. PMID 1389116
- [Background] Wiers RW, Gunning WB, Sergeant JA. Is a mild deficit in executive functions in boys related to childhood ADHD or to parental multigenerational alcoholism? J Abnorm Child Psychol. 1998 Dec;26(6):415-30. doi: 10.1023/a:1022643617017. PMID 9915649
- [Background] Willcutt EG, Doyle AE, Nigg JT, Faraone SV, Pennington BF. Validity of the executive function theory of attention-deficit/hyperactivity disorder: a meta-analytic review. Biol Psychiatry. 2005 Jun 1;57(11):1336-46. doi: 10.1016/j.biopsych.2005.02.006. PMID 15950006
- [Background] Schachar R, Tannock R, Marriott M, Logan G. Deficient inhibitory control in attention deficit hyperactivity disorder. J Abnorm Child Psychol. 1995 Aug;23(4):411-37. doi: 10.1007/BF01447206. PMID 7560554
- [Background] SWANSON IV, J. 2003. SNAP-IV Teacher and Parent Ratings Scale. Therapist's guide to learning and attention disorders, 487-500.
- [Background] ROID, G. H., & LEDBETTER, M. 2006. Wide range achievement test, fourth edition - progress monitoring version. Tampa, FL: Psychological Assessment Resources. disorder. Journal of Psychophysiology, 16, 97-106.
- [Background] Delis DC, Kaplan E, Kramer JH. Delis-Kaplan Executive Function System (D-KEFS): Examiner's manual. San Antonio, TX: The Psychological Corporation; 2001.
- [Background] GRODZINSKY, G. M. & DIAMOND, R. 1992. Frontal lobe functioning in boys with attention-deficit hyperactivity disorder. Developmental Neuropsychology, 8, 427-445.
- [Background] Mataro M, Garcia-Sanchez C, Junque C, Estevez-Gonzalez A, Pujol J. Magnetic resonance imaging measurement of the caudate nucleus in adolescents with attention-deficit hyperactivity disorder and its relationship with neuropsychological and behavioral measures. Arch Neurol. 1997 Aug;54(8):963-8. doi: 10.1001/archneur.1997.00550200027006. PMID 9267970
- [Background] Woodcock, R. W., McGrew, K. S., & Mather, N. (2001). Woodcock-Johnson tests of achievement III (WJ-III). Rolling Meadows, IL: Riverside Publishing.